CLINICAL TRIAL: NCT06991634
Title: An Open, Parallel Design Clinical Study to Evaluate the Pharmacokinetics and Safety of Azvudine Tablets in Healthy Adult Subjects and Healthy Elderly Subjects in Single and Multiple Doses
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of Azvudine Tablets in Healthy Adult Subjects and Healthy Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henan Genuine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-FNC-111
Record Dates: First submitted 2025-05-08; First posted 2025-05-28 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Azvudine; Pharmacokinetics; Safety
MeSH Terms: interventions — azvudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy adult subjects (Experimental)
  Interventions: Drug: Azvudine tablets
- Healthy elderly subjects (Experimental)
  Interventions: Drug: Azvudine tablets

INTERVENTIONS:
Drug: Azvudine tablets — Phase I: oral administration of 5 mg of Azvudine tablets on an empty stomach, single dose, 5 mg per dose.
  Phase II: oral administration of 5 mg of Azvudine tablets once a day on an empty stomach, 5 mg once a day, for 7 consecutive days.

SUMMARY:
Azvudine (FNC), a nucleoside reverse transcriptase inhibitor, make itself a better candidate to be co-formulated in other anti-HIV therapies, thus to improve patient's compliance. FNC is a broad-spectrum RNA virus inhibitor that inhibits the novel coronavirus RNA-dependent RNA polymerase (RdRp). This is an open, parallel design clinical study to evaluate the pharmacokinetics and safety of Azvudine tablets in healthy adult and elderly subjects in single and multiple doses. The study is divided into two stages. In the first stage, after a single oral administration of 5 mg of Azvudine tablets, biological sample collection and safety examination were performed. After completing the first phase of the test, the subjects can enter the second phase of the test after a 3-day washout period, and received oral administration of 5 mg Azvudine tablets once a day for 7 consecutive days, biological samples were collected and safety tests were performed.

ELIGIBILITY:
Inclusion Criteria:

Healthy adult subjects :

1. Age ≥ 18 years old and ≤ 45 years old, regardless of gender ;
2. Body mass index ( BMI ) in the range of 19.0-26.0 ( including the critical value ) ( BMI = weight ( kg ) / height 2 ( m2 ) ), male weight should be ≥ 50.0kg, female weight should be ≥ 45.0kg ;

Healthy elderly subjects :

1. Age ≥ 60 years old and ≤ 85 years old, regardless of gender ;
2. Body mass index ( BMI ) in the range of 18.0-35.0 ( including the critical value ) ( BMI = weight ( kg ) / height 2 ( m2 ) ) ;
3. Before the test, the existing disease if any was in a stable state and the treatment intervention or medication had no effect on this study.

Healthy adult subjects and healthy elderly subjects :

1. Patients who had no plan to become pregnant within 2 weeks before screening and 3 months after the end of the trial and agreed to take effective non-drug contraception during the trial ;
2. Understand and sign the informed consent.

Exclusion Criteria:

Healthy adult subjects:

1. The medical history, physical examination, laboratory items before the test, and the test-related examinations and test abnormalities have clinical significance, and the clinical research doctor judges that they are not eligible;
2. Subjects who have any history of prescription drugs, over-the-counter drugs, Chinese herbal medicines and healthcare products within 14 days before screening;

Healthy elderly subjects:

1. History or evidence of cardiovascular disease prior to screening: uncontrolled hypertension (SBP ≥ 170 mmHg and/or DBP ≥ 105 mmHg without antihypertensive therapy; SBP>160mmHg and/or DBP>100 mmHg with antihypertensive therapy), orthostatic hypotension, severe arrhythmias, heart failure, Adams-Stokes syndrome, unstable angina, history of myocardial infarction within 6 months prior to screening, tachycardia/bradycardia requiring medication, II-III degree atrioventricular block (excluding patients with pacemakers), or QTcF interval ≥ 450ms(Fridericia method);
2. The mini-mental state examination (MMSE) score results judged by the investigator are not suitable for this study;

Healthy adult subjects and healthy elderly subjects:

1. Allergic constitution, history of drug or food allergy, especially allergic to any ingredient in this product and accessories;
2. Patients with severe infection, trauma, or major surgery 4 weeks before screening, or who are scheduled to undergo surgery during the study;
3. Fever within 3 days before screening;
4. Those with serious diseases such as cerebral infarction and cancer in the past, except for benign diseases (such as liver cyst, renal cyst, fatty liver, etc.) based on chest radiograph and color Doppler ultrasound that do not need treatment;
5. Those who have participated in other clinical trials within 3 months before screening;
6. Drinking excessive amounts of tea, coffee and/or drinks rich in caffeine, xanthine and alcohol (more than 8 cups, 1 cup = 250mL) every day within 3 months before screening;
7. Smoking history within 12 months before screening (smoking number ≥ 5 cigarettes per day);
8. Those with a history of alcohol abuse within 12 months before screening (drinking ≥ 14 units of alcohol per week: 1 unit = 285mL of beer, or 25mL of spirits, or 150mL of wine) or those with a positive alcohol breath test (detection value> 0mg/100mL) before entering the group;
9. Those with a history of drug abuse within 12 months prior to screening or those who tested positive for addictive substances before entering the group;
10. Blood loss or blood donation ≥ 200mL within 8 weeks before screening (except for female physiological blood loss);
11. Pregnant and lactating women;
12. Those who cannot tolerate venipuncture blood collection and/or those who have a history of bleeding, acupuncture and/or blood collection vascular conditions are poor;
13. Those who have received the new coronavirus vaccine within 14 days before screening or other vaccines within 3 months before screening, or plan to receive the vaccine during the trial period;
14. The investigator considered it unsuitable to enter this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-08 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Plasma Concentration (Cmax) of Azvudine | Up to 36 hours post-dose.
Pharmacokinetics (PK): Area Under the Plasma Concentration Curve (AUC) of Azvudine | Up to 36 hours post-dose.
Pharmacokinetics (PK): Time to Maximum Plasma Concentration (Tmax) of Azvudine | Up to 36 hours post-dose.
Pharmacokinetics (PK): Elimination Half-life (T1/2) of Azvudine | Up to 36 hours post-dose.

SECONDARY OUTCOMES:
Occurrence of Adverse Events | From enrollment to the end of the study on Day 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Fifth Central Hospital, Tianjin, Tianjin Municipality, China